CLINICAL TRIAL: NCT00112294
Title: A Randomized Multicenter Phase III Study of Taxane/Carboplatin/Cetuximab Versus Taxane/Carboplatin as First-Line Treatment for Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Taxane/Carboplatin +/- Cetuximab as First-Line Treatment for Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-099
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; taxane; Docetaxel; Carboplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab+Taxane+Carboplatin (C/T/C) (Active Comparator): Cetuximab was administered at an initial dose (Week 1) of 400 mg/m^2 intravenous (IV) infusion (infused over 120 minutes) and a weekly maintenance dose of 250 mg/m^2 IV infusion (infused over 60 minutes). A cycle of therapy was defined as 3 weeks. Taxane was paclitaxel 225 mg/m^2 infused over 180 minutes on Day 1 and subsequently every 3 weeks or docetaxel 75 mg/m^2 infused over 60 minutes on Day 1 and subsequently every 3 weeks. Carboplatin was infused over 30 minutes on Day 1 and subsequently every 3 weeks.
  Interventions: Drug: Paclitaxel (Taxane); Drug: Docetaxel (Taxane); Drug: Carboplatin; Drug: Cetuximab
- Taxane+Carboplatin (T/C) (Active Comparator): A cycle of therapy was defined as 3 weeks. Taxane was paclitaxel 225 mg/m^2 infused over 180 minutes on Day 1 and subsequently every 3 weeks or docetaxel 75 mg/m^2 infused over 60 minutes on Day 1 and subsequently every 3 weeks. Carboplatin was infused over 30 minutes on Day 1 and subsequently every 3 weeks.
  Interventions: Drug: Paclitaxel (Taxane); Drug: Docetaxel (Taxane); Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel (Taxane) — IV, 225 mg/m^2
Drug: Docetaxel (Taxane) — IV, 75 mg/m^2
Drug: Carboplatin — AUC=6, q 3 weeks (6 cycles maximum)
Drug: Cetuximab — Intravenous, 400 mg/m^2, initial dose followed by 250 mg/m^2, weekly starting on Week 2
  Other Names: Erbitux
  Arms: Cetuximab+Taxane+Carboplatin (C/T/C)

SUMMARY:
The primary purpose of this clinical research study is to learn if patients treated with the combination of Taxane/Carboplatin plus Cetuximab (C/T/C) have a longer progression-free survival than patients treated with Taxane/Carboplatin (T/C) alone. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Must have advanced or metastatic non-small cell lung cancer that has not been previously treated with any chemotherapy.
* Tumor/disease lesions that can be measured bidimensionally.
* Must be able to carry-out work of light or sedentary nature (e.g. light house work, office work).
* Adequate recovery from recent surgery or radiation therapy.
* Must be at least 4 weeks from last major surgery or prior treatment with an investigational agent. At least 12 weeks from any radiation therapy to chest.
* Accessible for treatment, follow-up and required visits at a participating center(s).

Exclusion Criteria:

* Prior chemotherapy or adjuvant chemotherapy for the treatment of lung cancer.
* Prior treatment with cetuximab or other epidermal growth factor (EGFR)-targeted therapy.
* Prior severe infusion reaction to antibody therapy.
* Concurrent malignancy (previous malignancy without evidence of disease for 5 years will be allowed to enter trial).
* Concurrent chemotherapy or therapy with another investigational agent not indicated in the protocol.
* Serious uncontrolled medical disorders that would impair the ability to receive therapy.
* History of myocardial infarction within prior 3 months, uncontrolled angina, uncontrolled arrhythmia, or uncontrolled congestive heart failure.
* Symptomatic or uncontrolled metastases in the central nervous system. Subjects receiving a glucocorticoid for central nervous system (CNS) metastases are not eligible, but those receiving an anticonvulsant are eligible.
* Peripheral neuropathy >= grade 2 (Common Toxicity Criteria Adverse Event [CTCAE] Version 3.0).
* Inadequate hematologic and/or liver and/or kidney function.
* Sexually active and fertile individuals or partners of these individuals who are unwilling or unable to use an acceptable method of birth control for entire trial and up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment prior to study drug administration.
* Altered mental status or psychiatric condition that prohibits understanding or rendering of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (124):
- United States (124):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Anchorage, Alaska
  - Local Institution, Tucson, Arizona
  - Local Institution, Springdale, Arkansas
  - Local Institution, Anaheim, California
  - Local Institution, Bakersfield, California
  - Local Institution, Concord, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Gilroy, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Montebello, California
  - Local Institution, Oxnard, California
  - Local Institution, Rancho Mirage, California
  - Local Institution, San Diego, California
  - Local Institution, Stockton, California
  - Local Institution, Vista, California
  - Local Institution, Lakewood, Colorado
  - Local Institution, Binghamton, Connecticut
  - Local Institution, Hartford, Connecticut
  - Local Institution, New London, Connecticut
  - Local Institution, Norwich, Connecticut
  - Local Institution, Stamford, Connecticut
  - Local Institution, Waterbury, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Boca Raton, Florida
  - Local Institution, Boynton Beach, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Fort Myers, Florida
  - Local Institution, Inverness, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Lakeland, Florida
  - Local Institution, Lecanto, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Port Saint Lucie, Florida
  - Local Institution, Tamarac, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Augusta, Georgia
  - Local Institution, Columbus, Georgia
  - Local Institution, Marietta, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Evanston, Illinois
  - Local Institution, Joliet, Illinois
  - Local Institution, Naperville, Illinois
  - Local Institution, Normal, Illinois
  - Local Institution, Skokie, Illinois
  - Local Institution, Fort Wayne, Indiana
  - Local Institution, Muncie, Indiana
  - Local Institution, New Albany, Indiana
  - Local Institution, Terre Haute, Indiana
  - Local Institution, Vincennes, Indiana
  - Local Institution, Wichita, Kansas
  - Local Institution, Hazard, Kentucky
  - Local Institution, Paducah, Kentucky
  - Local Institution, Annapolis, Maryland
  - Local Institution, Baltimore, Maryland
  - Local Institution, Westminster, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Brockton, Massachusetts
  - Local Institution, Flint, Michigan
  - Local Institution, Free Soil, Michigan
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Jackson, Michigan
  - Local Institution, Dulluth, Minnesota
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Saint Louis Park, Minnesota
  - Local Institution, Jackson, Mississippi
  - Local Institution, Columbia, Missouri
  - Local Institution, Jefferson City, Missouri
  - Local Institution, Dover, New Hampshire
  - Local Institution, Newark, New Jersey
  - Local Institution, Cooperstown, New York
  - Local Institution, New City, New York
  - Local Institution, New Rochelle, New York
  - Local Institution, Northport, New York
  - Local Institution, Rochester, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Valhalla, New York
  - Local Institution, Burlington, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Gastonia, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Greenville, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Morganton, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Bismarck, North Dakota
  - Local Institution, Canton, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Dayton, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Bethlehem, Pennsylvania
  - Local Institution, Dunmore, Pennsylvania
  - Local Institution, Harrisburg, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pottstown, Pennsylvania
  - Local Institution, Sayre, Pennsylvania
  - Local Institution, West Reading, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Columbia, South Carolina
  - Local Institution, Mt. Pleasant, South Carolina
  - Local Institution, Spartanburg, South Carolina
  - Local Institution, Sumter, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Collierville, Tennessee
  - Local Institution, Cookeville, Tennessee
  - Local Institution, Amarillo, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Lubbock, Texas
  - Local Institution, Danville, Virginia
  - Local Institution, Lynchburg, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Everett, Washington
  - Local Institution, Lacey, Washington
  - Local Institution, Tacoma, Washington
  - Local Institution, Huntington, West Virginia
  - Local Institution, La Crosse, Wisconsin
  - Local Institution, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 755 participants were enrolled and 676 were randomized into the study. 79 participants were not randomized (6 deaths; 1 lost to follow up; 1 poor/non-compliance; 49 no longer met study criteria; 17 participant request; 2 required concurrent radiation; 1 insurance issue; 1 doctor discretion; 1 unknown).
Groups:
- Cetuximab+Taxane+Carboplatin (C/T/C): Cetuximab was administered at an initial dose (Week 1) of 400 mg/m^2 IV infusion (infused over 120 minutes) and a weekly maintenance dose of 250 mg/m^2 IV infusion (infused over 60 minutes). A cycle of therapy was defined as 3 weeks. Taxane was paclitaxel 225 mg/m^2 infused over 180 minutes on Day 1 and subsequently every 3 weeks or docetaxel 75 mg/m^2 infused over 60 minutes on Day 1 and subsequently every 3 weeks. Carboplatin was infused over 30 minutes on Day 1 and subsequently every 3 weeks.
Period: Overall Study
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Started | 325 (338 randomized and 325 treated.) | 320 (338 randomized and 320 treated.)
Never Treated | 13 (Number by randomized group = 11, but 2 participants received C/T/C instead of T/C.) | 18 (Number by randomized group = 20, but 2 participants received C/T/C instead of T/C.)
Completed | 320 (Off all study therapies.) | 320 (Off all study therapies.)
Not Completed | 5 | 0
Not completed — Still on study | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C) | Total
Number analyzed (Participants) | 338 | 338 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.0) | 63.9 (10.3) | 64.0 (10.2)
Age, Customized [Number; unit: participants]
  <65 years | 171 | 165 | 336
  >= 65 years | 167 | 173 | 340
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 134 | 280
  Male | 192 | 204 | 396
Race/Ethnicity, Customized [Number; unit: Participants] — 'Other race' includes 1 American Indian or Alaska native and 3 native Hawaiian or other pacific islander.
  Participants
    Asian | 6 | 10 | 16
    Black | 25 | 24 | 49
    White | 296 | 300 | 596
    Other race | 11 | 4 | 15
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: Participants] — The ECOG PS is used to assess disease severity. A score of 0 is fully active; 1 is restricted physically strenuous activity; 2 is ambulatory but unable to work; 3 is capable of only limited self care; 4 is completely disabled; 5 is dead. Missing includes participants whose pre-treatment PS > 14 days prior to first dose.
  Participants
    0=fully active | 110 | 114 | 224
    1=restricted physically strenuous activity | 221 | 220 | 441
    2=ambulatory but unable to work | 4 | 2 | 6
    3=capable of only limited self care | 0 | 1 | 1
    4=completely disabled | 0 | 0 | 0
    5=dead | 0 | 0 | 0
    Missing | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kg] — 3 participants in the C/T/C group did not have values for this measure. 1 participant in the C/T group did not have a value for this measure.
  kg | 75.0 (17.1) | 75.3 (18.1) | 75.1 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Months of Progression-free Survival (PFS)
Description: Interval between randomization date & earliest date of disease progression/death due to any cause, assessed by the Independent Radiology Review Committee (IRRC) using modified World Health Organization (WHO) criteria to define progressive disease (PD): >=25% increase in sum of products of diameters (SOPD) of lesions compared with smallest SOPD recorded for study period or progression of any non-index lesion/appearance of new lesion. If no progression/death, date of last tumor assessment used. For participants who had no on-study tumor assessments & were still alive, date of randomization used.
Time Frame: From randomization to evidence of disease progression/death or date of last tumor assessment (up to 26 months).
Population: All randomized participants (intention to treat population).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 338 | 338
Months | 4.40 [4.11 to 5.06] | 4.24 [3.94 to 4.63]
Statistical Analysis 1: Comparison: Cetuximab+Taxane+Carboplatin (C/T/C) vs Taxane+Carboplatin (T/C); Confidence intervals calculated using Brookmeyer and Crowley method. Primary analysis was comparison of PFS between arms performed by 2-sided alpha=0.05 level, log-rank test, stratified by ECOG PS (0/1) and intended on-study taxane (docetaxel or paclitaxel). Null hypothesis was that PFS was equal in both groups. Power calculations indicated that >=510 events (IRRC progressions/deaths) would lead to >=90% power at the 5% level for rejecting the null hypothesis, given a true hazard ratio of 0.75; Test type: Superiority or Other; p = 0.2358, Log Rank — Since only 1 primary comparison was conducted, no adjustment for multiple comparisons was needed; Hazard Ratio (HR) = 0.902, 95% CI 2-sided [0.761 to 1.069] — The hazard ratio of C/T/C to T/C was estimated by means of a stratified Cox's proportional hazard model, with treatment as the single covariate

2. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: Tumor response was defined as the number of participants whose best response was CR or PR, per the IRRC assessment, using the modified WHO criteria: CR: disappearance of all index/non-index lesions; PR: >= 50% reduction in the SOPD of index lesions compared with the baseline SOPD, with no evidence of progression. To qualify as CR or PR, no new lesions could be present.
Time Frame: From randomization to end of study drug therapy (up to 174 weeks).
Population: All randomized participants (intention to treat population).
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 338 | 338
Participants | 87 | 58
Statistical Analysis 1: Comparison: Cetuximab+Taxane+Carboplatin (C/T/C) vs Taxane+Carboplatin (T/C); The 2 groups were compared by means of a Cochran-Mantel-Haenszel (CMH) (alpha = 0.05 level) test stratified by ECOG PS (0 or 1) and intended on-study taxane (paclitaxel, docetaxel), as recorded at the time of randomization; Test type: Superiority or Other; p = 0.0066, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.675, 95% CI 2-sided [1.152 to 2.436] — The odds ratio is presented for C/T/C to T/C

3. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Disease control was defined as the number of participants whose best response was CR, PR, or SD, per the IRRC assessment, using the modified WHO criteria: CR: disappearance of all index/non-index lesions; PR:>= 50% reduction in the SOPD of index lesions compared with the baseline SOPD, with no evidence of progression (to qualify as CR or PR, no new lesions could be present); SD: participants who did not meet the criteria for CR, PR, or PD (PD:>=25% increase in SOPD of lesions compared with smallest SOPD recorded for study period or progression of any non-index lesion/appearance of new lesion).
Time Frame: From randomization to end of study drug therapy (up to 174 weeks).
Population: All randomized participants (intention to treat population).
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 338 | 338
Participants | 230 | 212
Statistical Analysis 1: Comparison: Cetuximab+Taxane+Carboplatin (C/T/C) vs Taxane+Carboplatin (T/C); The 2 groups were compared by means of a CMH (alpha = 0.05 level) test stratified by ECOG PS (0 or 1) and intended on-study taxane (paclitaxel, docetaxel), as recorded at the time of randomization; Test type: Superiority or Other; p = 0.1501, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.265, 95% CI 2-sided [0.918 to 1.741] — The odds ratio is presented for C/T/C to T/C

4. Secondary Outcome: Median Number of Months of Response
Description: Median number of months of response (time from first occurrence of CR/PR to date of PD/death, [per IRRC assessment,using modified WHO criteria]) calculated for participants whose best response=CR/PR.For participants who did not progress/die, date of last tumor assessment used.CR:disappearance of all index/non-index lesions;PR:>= 50% reduction in SOPD of index lesions compared with baseline, no evidence of progression.No new lesions present.PD:>=25% increase in SOPD of lesions compared with smallest SOPD recorded for study period or progression of any non-index lesion/appearance of new lesion.
Time Frame: Time from first occurrence of CR or PR (whichever was recorded first) to the date of PD, death or date of last tumor assessment (up to 19 months).
Population: All randomized participants with a best response of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 87 | 58
Months | 5.55 [4.40 to 6.83] | 4.90 [4.24 to 5.72]

5. Secondary Outcome: Median Number of Months to Response
Description: The median number of months to response was calculated for participants whose best response was CR or PR. It was defined as the time from the first dose of study therapy to the first date that criteria for PR or CR (whichever occurred first)were met. Response was assessed by the IRRC, using the modified WHO criteria: CR: disappearance of all index/non-index lesions; PR: >= 50% reduction in the SOPD of index lesions compared with the baseline SOPD, with no evidence of progression. To qualify as CR or PR, no new lesions could be present.
Time Frame: Time from first dose of study therapy to the date of PR or CR, whichever occurred first (up to 13 months).
Population: All randomized participants with a best response of CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 87 | 58
Months | 1.38 [1.08 to 12.65] | 1.35 [0.99 to 4.83]

6. Secondary Outcome: Median Number of Months of Survival
Description: The median number of months of survival was defined as the time from randomization to the date of death. For participants who did not die, the date of last contact was used.
Time Frame: From randomization to death or date of last contact (up to 41 months).
Population: All randomized participants (intention to treat population).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 338 | 338
Months | 9.69 [8.28 to 11.50] | 8.38 [7.33 to 9.92]
Statistical Analysis 1: Comparison: Cetuximab+Taxane+Carboplatin (C/T/C) vs Taxane+Carboplatin (T/C); Confidence intervals were calculated using Brookmeyer and Crowley method. Analysis was a comparison of survival between groups by means of a 2-sided, alpha=0.05 level, log-rank test, stratified by ECOG PS (0/1) and intended on-study taxane (docetaxel or paclitaxel). Null hypothesis was that survival was equal in both treatment arms. Power calculations indicated that >= 558 events would lead to at >=75% power at the 5% level for rejecting the null hypothesis, given a true hazard ratio of 0.8; Test type: Superiority or Other; p = 0.1685, Log Rank — An interim analysis on survival was performed. Final p-value was adjusted using an alpha spending function. At the interim analysis (data not reported here) the type 1 error was 0.0001, and the rest is for the final look; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.754 to 1.051] — The hazard ratio of C/T/C to T/C was estimated by means of a stratified Cox's proportional hazard model with treatment as the single covariate

7. Secondary Outcome: Number of Participants With Improvement of Symptoms
Description: Symptoms were assessed using the Functional Assessment of Cancer Therapy - Lung Cancer Subscale (FACT-LCS) questionnaire. This 7-item scale has scores ranging from 0 (severely symptomatic in all symptoms assessed) to 28 (symptom-free on all symptoms assessed). Symptom response (improvement) was defined as >= 2-point increase from baseline in score (maintained for 2 consecutive assessments, at least 3 weeks apart). Participants with a baseline score of >= 27 were not evaluable, as it would not have been possible to show an improvement. Participants with no baseline data were also not evaluable.
Time Frame: From randomization to evidence of disease progression/death or date of last symptom assessment (up to 33 weeks).
Population: All randomized participants who completed a baseline FACT-LCS questionnaire (ie, who completed a questionnaire <=14 days prior to treatment, or if they were never treated, <=14 days prior to randomization) and who had a baseline score of 26 or less.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 328 | 323
Participants | 107 | 92
Statistical Analysis 1: Comparison: Cetuximab+Taxane+Carboplatin (C/T/C) vs Taxane+Carboplatin (T/C); Improvement of symptoms was compared between groups by means of a CMH (alpha = 0.05 level) test stratified by ECOG PS (0 or 1) and intended on-study taxane (paclitaxel, docetaxel), as recorded at the time of randomization; Test type: Superiority or Other; p = 0.26, Cochran-Mantel-Haenszel

8. Secondary Outcome: Median Number of Months Until Symptomatic Progression (Worsening of Symptoms)
Description: Symptoms were assessed using the FACT-LCS questionnaire. This 7-item scale has scores ranging from 0 (severely symptomatic) to 28 (symptom-free). Symptomatic progression was defined as >= 2-point decrease from baseline in score (maintained for 2 consecutive assessments at least 3 weeks apart). Time to symptomatic progression was defined as the time from randomization to date of symptoms worsening. For participants with no symptom progression, the date of the last symptom assessment was used. See also Outcome Measure 15.
Time Frame: From randomization to evidence of disease progression/death or date of last symptom assessment (up to 33 weeks).
Population: All randomized participants who completed baseline FACT-LCS questionnaire (ie, completed questionnaire <=14 days prior to treatment, or if they were never treated, <=14 days prior to randomization) and who had a baseline score greater than or equal to 2. As the median was not reached, no data are presented here (see Outcome Measure 15).
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Died, or Experienced Other Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). An SAE was defined as an AE that resulted in death, was life-threatening, required hospitalization (or prolongation of existing hospitalization), or was an important medical event.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants. The AEs represented here include SAEs, which are not included in the AE count represented in the AE xml upload section. As such, these numbers may not match.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants
  Death | 38 | 27
  Serious adverse events | 183 | 121
  Adverse events | 324 | 320

10. Secondary Outcome: Number of Participants Experiencing AEs Leading to Study Drug Discontinuation
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). The results presented are stratified according to which drug was discontinued.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
participants
  Cetuximab | 100 | 0
  Taxane | 80 | 54
  Carboplatin | 78 | 52

11. Secondary Outcome: Number of Participants Experiencing Other Significant AEs: Acneform Rash
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). For this study, it was decided that AEs that were categorized under the composite term "acneform rash" were of particular importance. These AEs were: rash, rash pustular, rash erythematous, dermatitis acneiform, dermatitis exfoliative, rash papular, rash pruritic, rash generalised, rash macular, rash maculo-papular, acne, acne pustular, skin desquamation and dry skin.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants | 246 | 56

12. Secondary Outcome: Number of Participants Experiencing Other Significant AEs: Infusion Reaction
Description: AE=any new untoward medical occurrence or worsening of pre-existing medical condition (even if not caused by the study drug). For this study, it was decided that AEs that were categorized under the composite term "infusion reaction" were of particular importance. These AEs were: infusion-related reaction, hypersensitivity, anaphylactic reaction, anaphylactic shock, and anaphylactoid reaction regardless of when they occurred. The terms dyspnea, pyrexia and chills were also grouped under infusion reaction, provided the onset date of these toxicities occurred on the first day of study treatment.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants | 45 | 18

13. Secondary Outcome: Number of Participants Experiencing Other Significant AEs: Cardiac AEs
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). For this study, it was decided that AEs that were categorized under the composite term "cardiac AE" were of particular importance. These AEs, coded as preferred or other level Medical Dictionary for Regulatory Activities [MedDRA] terms were: coronary artery disorders, cardiac arrhythmias, heart failures not elsewhere classified, left ventricular failures, sudden cardiac death, cardiac death and sudden death.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants | 58 | 25

14. Secondary Outcome: Number of Participants Who Exprienced the Most Frequent Grade 3-4 Hematology Abnormalities Occurring in >=5% Participants
Description: Abnormalities were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 3.0. The scale is graded from 1 (least severe) to 4 (life threatening). Grade 3 and 4 criteria are defined as follows: Neutropenia: Grade 3, neutrophils <1.0 - 0.5 x 10^9/L; Grade 4, <0.5 x 10^9/L. Leukopenia: Grade 3, leukocytes <2.0 - 1.0 x 10^9/L; Grade 4, <1.0 x 10^9/L. Thrombocytopenia: Grade 3, platelets <50.0 - 25.0 x 10^9/L; Grade 4, <25.0 x 10^9/L. Anemia: Grade 3, hemoglobin <4.9 - 4.0 millimoles (mmol)/L, Grade 4, <4.0 mmol/L.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants
  Neutropenia | 198 | 177
  Leukopenia | 139 | 97
  Thrombocytopenia | 33 | 29
  Anemia | 17 | 15

15. Other Pre Specified Outcome: Median Change From Baseline in Symptoms, by Time Point
Description: Symptoms were assessed using the FACT-LCS questionnaire. This 7-item scale has scores ranging from 0 (severely symptomatic) to 28 (symptom-free). The median change from baseline score was calculated at 3-weekly intervals. See also Outcome Measure 8.
Time Frame: From randomization to evidence of disease progression/death or date of last symptom assessment (up to 33 weeks).
Population: All randomized participants who completed a baseline FACT-LCS questionnaire (ie, completed questionnaire <=14 days prior to treatment, or if they were never treated, <=14 days prior to randomization). n = number of participants with a score at both the baseline and at the specified time point (each arm respectively).
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 336 | 335
Units on a scale
  3 weeks (n = 286, 257) | 1.0 [-1.0 to 3.0] | 0.8 [-2.0 to 3.0]
  6 weeks (n = 254, 221) | 1.0 [-2.0 to 4.0] | 1.0 [-2.0 to 4.0]
  9 weeks (n = 203, 175) | 1.0 [-2.0 to 4.0] | 1.0 [-2.0 to 4.0]
  12 weeks (n = 178, 161) | 1.0 [-2.0 to 4.0] | 0.0 [-2.0 to 4.0]
  15 weeks (n = 155, 121) | 1.0 [-2.0 to 4.0] | 1.0 [-2.0 to 5.0]
  18 weeks (n = 126, 91) | 1.0 [-1.0 to 4.0] | 2.0 [-2.0 to 5.0]
  21 weeks (n = 96, 43) | 2.0 [-1.0 to 4.0] | 3.0 [-1.0 to 7.0]
  24 weeks (n = 90, 41) | 2.0 [-2.0 to 5.0] | 1.0 [-1.0 to 5.0]
  27 weeks (n = 60, 22) | 3.0 [-1.0 to 5.0] | 3.5 [-1.0 to 7.0]
  30 weeks (n = 56, 15) | 1.5 [-1.0 to 5.0] | 3.0 [0.0 to 5.0]
  33 weeks (n = 43, 7) | 2.1 [-1.0 to 6.0] | 3.0 [-1.0 to 8.0]

16. Secondary Outcome: Number of Participants Who Experienced the Most Frequent Grade 3-4 Serum Chemistry Abnormalities Occurring in >=5% Participants
Description: Abnormalities were graded according to the NCI CTC, version 3.0. The scale is graded from 1 (least severe) to 4 (life threatening). Grade 3 and 4 criteria are defined as follows: Hyperglycemia (non-fasting): Grade 3, serum glucose >13.9 - 27.8 mmol/L; Grade 4 >27.8 mmol/L or acidosis. Hypomagnesemia: Grade 3, serum magnesium >1.23 - 3.30 mmol/L; Grade 4 >3.30 mmol/L. Hyponatremia: Grade 3, serum sodium <130 - 120 mmol/L; Grade 4 <120 mmol/L. Low albumin: Grade 3, serum albumin <20 g/L; Grade 4 not applicable.
Time Frame: From start of study drug therapy up to 30 days after the last dose (up to 178 weeks).
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 325 | 320
Participants
  Hyperglycemia (non-fasting) | 33 | 36
  Hypomagnesemia | 26 | 2
  Hyponatremia | 25 | 21
  Low albumin | 17 | 9

17. Secondary Outcome: Number of Participants Who Had Unscheduled Visits to Physicians, Clinics, Hospitals and Other Unscheduled Major Medicinal Procedures
Description: Participants were to complete log to collect information on unscheduled visits to physicians,clinics,hospitals & other unscheduled major procedures.If asked, participants were to complete and return log to site upon routinely scheduled visits.The purpose of this exploratory analysis was to understand the economical implications as a secondary objective.This was not a pivotal study & therefore not needed to support any arguments with regulatory authorities concerning cost-benefit,hence,it was not necessary to conduct this analysis. There is no intent on conducting this analysis in the future.
Time Frame: Day 1 of each cycle of treatment, at the end of study therapy evaluation and at the first follow-up visit (6 weeks after the end of study therapy evaluation).
Population: This analysis was not performed.
Arm/Group | Cetuximab+Taxane+Carboplatin (C/T/C) | Taxane+Carboplatin (T/C)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The AEs represented here do not include SAEs. As such, these numbers may not match with the AEs presented as an Outcome Measure.
Arm/Group | Cetuximab+Taxane+Carboplatin | Taxane+Carboplatin
Serious Adverse Events (participants affected / at risk) | 183/325 | 121/320
Other Adverse Events (participants affected / at risk) | 322/325 | 317/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab+Taxane+Carboplatin (N=325) | Taxane+Carboplatin (N=320)
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Asthenia (General disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 6 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 3
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cellulitis (Infections and infestations) | 3 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 3
Cerebrovascular accident (Nervous system disorders) | 5 | 4
Cervical cord compression (Nervous system disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Clostridial infection (Infections and infestations) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Convulsion (Nervous system disorders) | 4 | 2
Deep vein thrombosis (Vascular disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 24 | 11
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 8
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 11 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Ileus (Gastrointestinal disorders) | 2 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Infection (Infections and infestations) | 2 | 3
Infective myositis (Infections and infestations) | 0 | 1
Infusion related reaction (General disorders) | 2 | 0
International normalised ratio increased (Investigations) | 1 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung infection (Infections and infestations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 11
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 4
Nephritis (Renal and urinary disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 9 | 4
Neutropenic infection (Infections and infestations) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 3
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pain (General disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 4 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pneumonia (Infections and infestations) | 18 | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 2
Renal pain (Renal and urinary disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Sepsis (Infections and infestations) | 6 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 4 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 5
Syncope vasovagal (Nervous system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombosis (Vascular disorders) | 3 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 1 | 1
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5
Vomiting projectile (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab+Taxane+Carboplatin (N=325) | Taxane+Carboplatin (N=320)
Abdominal pain (Gastrointestinal disorders) | 40 | 27
Alopecia (Skin and subcutaneous tissue disorders) | 118 | 141
Anaemia (Blood and lymphatic system disorders) | 26 | 26
Anorexia (Metabolism and nutrition disorders) | 131 | 97
Anxiety (Psychiatric disorders) | 32 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 | 51
Asthenia (General disorders) | 36 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 41
Bone pain (Musculoskeletal and connective tissue disorders) | 25 | 25
Chills (General disorders) | 25 | 22
Confusional state (Psychiatric disorders) | 16 | 16
Constipation (Gastrointestinal disorders) | 147 | 99
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 81
Decreased appetite (Metabolism and nutrition disorders) | 28 | 20
Dehydration (Metabolism and nutrition disorders) | 79 | 46
Depression (Psychiatric disorders) | 38 | 28
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 58 | 2
Diarrhoea (Gastrointestinal disorders) | 156 | 105
Dizziness (Nervous system disorders) | 67 | 47
Dry mouth (Gastrointestinal disorders) | 18 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 68 | 11
Dysgeusia (Nervous system disorders) | 60 | 46
Dyspepsia (Gastrointestinal disorders) | 48 | 29
Dysphagia (Gastrointestinal disorders) | 22 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 106 | 104
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 | 18
Exfoliative rash (Skin and subcutaneous tissue disorders) | 26 | 1
Fatigue (General disorders) | 243 | 228
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 | 19
Headache (Nervous system disorders) | 36 | 33
Hypersensitivity (Immune system disorders) | 22 | 8
Hypoaesthesia (Nervous system disorders) | 20 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 31 | 2
Hypotension (Vascular disorders) | 36 | 19
Insomnia (Psychiatric disorders) | 86 | 69
Localised infection (Infections and infestations) | 19 | 0
Mucosal inflammation (General disorders) | 50 | 19
Muscular weakness (Musculoskeletal and connective tissue disorders) | 29 | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 25 | 26
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 45 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 36
Nail disorder (Skin and subcutaneous tissue disorders) | 17 | 5
Nausea (Gastrointestinal disorders) | 198 | 161
Neuropathy peripheral (Nervous system disorders) | 61 | 64
Neutropenia (Blood and lymphatic system disorders) | 29 | 19
Non-cardiac chest pain (General disorders) | 31 | 29
Oedema peripheral (General disorders) | 55 | 46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 34
Paraesthesia (Nervous system disorders) | 19 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 43 | 51
Pruritus (Skin and subcutaneous tissue disorders) | 45 | 17
Pyrexia (General disorders) | 43 | 31
Rash (Skin and subcutaneous tissue disorders) | 186 | 47
Stomatitis (Gastrointestinal disorders) | 72 | 41
Tachycardia (Cardiac disorders) | 24 | 6
Upper respiratory tract infection (Infections and infestations) | 22 | 13
Urinary tract infection (Infections and infestations) | 26 | 13
Vision blurred (Eye disorders) | 21 | 11
Vomiting (Gastrointestinal disorders) | 107 | 93
Weight decreased (Investigations) | 67 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.